CLINICAL TRIAL: NCT06079606
Title: The Effects of Antibiotic Exposure in Early Infancy on Vaccine Responses
Status: Active, not recruiting | Type: Observational
Sponsor: Landspitali University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: e-INFANT-2
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Immune Responses; Antibiotic Treatment
Keywords: Antibiotics; Immune Responses; Vaccinations; Children; Rotavirus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and salivary samples collected for measurement of immune responses. Stool samples collected for microbiome analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: Term children born with caesarean section (their mothers received intra-operative antibiotics)
  Interventions: Other: Antibiotic treatment
- Group B: Term vaginally born children and their mothers received intra-partum antibiotics
  Interventions: Other: Antibiotic treatment
- Group C: Term vaginally born children that received systemic antibiotics during the first week of life for at least 48 hours
  Interventions: Other: Antibiotic treatment
- Group D (Control group): Term vaginally born children that had not received systemic antibiotics at the time of recruitment

INTERVENTIONS:
Other: Antibiotic treatment — Children will be assigned to groups according to antibiotic exposure in early life. No antibiotics will be given in the study.
  Groups: Group A; Group B; Group C

SUMMARY:
This prospective cohort study will include 200 term children born in Landspitali University Hospital in Iceland. The cohort will be divided into four groups according to antibiotic exposure of which one is the control group. Children's immune responses to live oral rotavirus vaccine as well as conventional vaccinations given at three, five and 12 months old will be determined by measuring salivary and serologic responses. Responses will be compared between the four groups. Stool samples will also be collected from participants and the composition of the microbiome compared between the four groups.

DETAILED DESCRIPTION:
This prospective cohort study will evaluate the development of the immune system by means of evaluating the immune responses to oral rotavirus vaccine and the scheduled childhood vaccinations in Iceland, at the age of three, five and 12 months, in four different groups of term children born in Iceland.

The cohort will be divided into the following groups:

* Group A: Term children born with elective caesarean section (their mothers received intra-operative antibiotics).
* Group B: Term vaginally born children and their mothers received intra-partum antibiotics.
* Group C: Term vaginally born children that received systemic antibiotics during the first week of life for at least 48 hours.
* Group D: Term vaginally born children that had not received systemic antibiotics at the time of recruitment.

Parents of children born with elective caesarean section in Landspitali or born vaginally and their mothers received intra-partum antibiotics as well as parents of children in the Neonatal Intensive Care Unit receiving systemic antibiotics during the first week of life will be offered to take part in the study (Groups A, B and C). Parents of children coming to a five day old check up at the Children's Hospital in Landspitali will also be offered to take part in the study (Group D). Sample size calculations show that to detect a 30% difference in immune responses to vaccines with 80% power, 40 infants are needed for analysis in each group. To account for late exclusions due to antibiotic use or drop-out due to other reasons, 50 infants will be recruited to each group. Participants will receive vaccination with the oral live attenuated rotavirus vaccine, Rotarix, at six weeks old and again at three months old. Participants will receive vaccinations with Pentavac against diphtheria, tetanus, pertussis, haemophilus influenza type B and polio and Synflorix against pneumococci at their Health Care Centre according to scheduled childhood vaccinations in Iceland at three, five and 12 months old. Salivary and blood samples will be taken from participants just before the first vaccination with Rotarix at six weeks old and again at six months (four weeks after the second dose of Pentavac and Synflorix) and at 13 months old (four weeks after the third dose of Pentavac and Synflorix). Specific antibody levels against rotavirus, pertussis, diphtheria, tetanus, haemophilus influenzae type B, polio virus and pneumococci will be measured. Parents of participants will be given two stool sample kits and asked to take one from their child at six weeks old (before the first dose of rotavirus vaccine) and then another at three months old. In case of detection of differences in antibody response, these samples will be sent for microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* All term children born in Iceland from 2022-2023

Exclusion Criteria:

* Children born with emergency caesarean section
* Children born before 36 weeks of gestation
* Children diagnosed with primary or secondary immunodeficiency
* Use of immunosuppressive drugs at recruitment or during the follow up period (excluding inhaled corticosteroids and short term oral corticosteroids (<3 consecutive days).
* Children with chromosomal, genetic or other congenital diseases or abnormalities
* Children with severe, chronic diseases or disabilities
* Informed consent not signed by parents

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Group A: In total 50 term children born in Iceland during the time period 2022-2023, delivered with elective caesarean section (their mothers received intra-operative antibiotics).
  * Group B: In total 50 term children born in Iceland during the time period 2022-2023, delivered vaginally and their mothers received intra-partum antibiotics.
  * Group C: In total 50 term children born in Iceland during the time period 2022-2023, delivered vaginally and received systemic antibiotics during the first week of life for at least 48 hours.
  * Control group (Group D): In total 50 term children born in Iceland during the time period 2022-2023, delivered vaginally and received no systemic antibiotics at the time of recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum antibody response to rotavirus | 2 years
  Serum IgA against rotavirus
Salivary antibody response to rotavirus | 2 years
  Salivary IgA levels against rotavirus
Serum antibody response to other microbes | 2 years
  Serum IgG against other microbes
Salivary antibody response to other microbes | 2 years
  Salivary IgG against other microbes

SECONDARY OUTCOMES:
Composition of the microbiome | 3 years
  16s rRNA analysis of stool microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- Landspitali University Hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No